CLINICAL TRIAL: NCT05840757
Title: Non-Invasive MOnitoring in Transcathether Aortic Valve Implantation - A Single-center, Prospective, Interventional Study With the ClearSight® Finger Cuff
Brief Title: Non-Invasive MOnitoring in Transcathether Aortic Valve Implantation
Acronym: NIMO-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Thomas Nestelberger, Head of Structural Cardiology, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Basel
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Aortic Valve Disease
Keywords: Transcatheter aortic valve implantation; hemodynamic parameter
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodynamic Monitoring (Other): Simultaneous measurement of hemodynamic parameters such as Cardiac output, cardiac index and blood pressure with invasive right heart catheterization and non-invasive application of the Clearsight Finger Cuff.
  Interventions: Device: HemoSphere ClearSight Module

INTERVENTIONS:
Device: HemoSphere ClearSight Module — The Clear Sight system consists of a finger cuff connected to a monitor It will be applied to the patients finger before and removed after the TAVI procedure.

SUMMARY:
In patients with severe aortic stenosis (AS) undergoing transcatheter aortic valve implantation (TAVI) minimal evidence is available for invasive hemodynamic monitoring and no evidence for tools able to measure traditionally invasive parameters non-invasively for peri-procedural guidance and post-interventional management.

The aim of this study is to evaluate the effectiveness and safety of a non-invasive hemodynamics monitoring tool called ClearSight for monitoring during TAVI procedures compared with standard invasive measurements.

DETAILED DESCRIPTION:
In patients with severe aortic stenosis (AS) undergoing transcatheter aortic valve implantation (TAVI) minimal evidence is available for invasive hemodynamic monitoring and no evidence for tools able to measure traditionally invasive parameters non-invasively for peri-procedural guidance and post-interventional management.

The aim of this study is to evaluate the effectiveness and safety of a non-invasive hemodynamics monitoring tool called ClearSight for monitoring during TAVI procedures compared with standard invasive measurements.

The ClearSight monitoring system works non-invasively by utilizing an inflatable finger cuff which adjusts automatically to measure the arterial blood pressure which enables the calculation of parameters such as cardiac output or index. Multiple studies have demonstrated the reliability and feasibility of continuous non-invasive monitoring, in different settings, however it was never performed in patients undergoing TAVI.

The ClearSight monitoring system will be directly compared to invasive measurements of hemodynamic parameters during the procedure. In addition, information regarding baseline hemodynamics and its changes during/after procedure may give important information on peri- and post-procedural management and short-term outcomes and discharge planning. A tool, providing this information non-invasively with the same accuracy might result in a major improvement in daily practice..

ELIGIBILITY:
Inclusion Criteria:

• Adult patients (>18 years old) with severe aortic stenosis undergoing elective TAVI.

Exclusion Criteria:

* Emergency indication for TAVI
* Severe tricuspid regurgitation
* Severe mitral stenosis or severe regurgitation
* Invasive right heart catheterization impossible
* Dependency on right ventricle pacing immediately after TAVI implantation
* Vulnerable subjects
* Known or suspected non-compliance, drug or alcohol abuse
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation affecting this study
* Previous enrolment into the current investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | During aortic valve implantation which generally takes about 40mins
  Cardiac Output (CO in L/min)
Cardiac Index | During aortic valve implantation which generally takes about 40mins
  Cardiac Index (CI in L/min/m2)
Systolic blood pressure | During aortic valve implantation which generally takes about 40mins
  systolic blood pressure (sBP in mmHg)
Diastolic blood pressure | During aortic valve implantation which generally takes about 40mins
  diastolic blood pressure (dBP in mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No